CLINICAL TRIAL: NCT06416007
Title: A Phase 2 Study of Lattice Radiotherapy for Dose-Escalated Palliation of Bulky Tumors
Brief Title: Lattice Radiotherapy for Dose-Escalated Palliation of Bulky Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Andrew Frankart, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-RT-23-01
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Metastatic Cancer; Locally Advanced; Locally Advanced Solid Tumor; Locally Advanced Carcinoma
Keywords: Radiation; Radiotherapy; Bulky; Spatial fractionation; Lattice therapy; Palliative; Palliation
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lattice radiation therapy (LRT) (Experimental): Lattice radiation therapy (LRT) : 5 fractions
  Interventions: Radiation: Lattice therapy (LRT)

INTERVENTIONS:
Radiation: Lattice therapy (LRT) — 5 Fractions LRT

SUMMARY:
The purpose of this research study is to determine if lattice radiation therapy (LRT) will provide better treatment for bulky (large) tumors than current standard of care radiotherapy.

DETAILED DESCRIPTION:
This will be a single-institution, single-arm Phase II trial with an anticipated total of 37 patients enrolled. Treatment will consist of 5 fractions of lattice radiation therapy delivered every other day. The primary endpoints will include the efficacy of lattice therapy as evaluated by ORR (CR or PR per RECIST criteria) at 60 days (2 months) post-treatment and safety. Toxicity will be evaluated at day 5 (+/- 2 days), day 15 (+/- 5 days), day 30 (+/- 5 days), and day 60 (+/- 7 days) post-completion of lattice therapy. This study will also include a translational analysis of the impact of lattice therapy on systemic immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor malignancy with a clinical indication for radiation
* Patients must have measurable disease
* Target lesion(s) which are amenable to lattice therapy plan
* When applicable, target lesion for radiation amenable to immobilization during delivery of radiotherapy
* Age ≥18 years.
* ECOG Performance status ≤2
* Life expectancy greater than 3 months
* Women of child-bearing potential and men must agree to avoid conception via abstinence (ideal) or a method of birth control (e.g., hormonal or barrier method of birth control) prior to study entry and for at least 30 days after completion of lattice therapy administration.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients receiving cytotoxic chemotherapy or known radiosensitizing agents within 5 days before or after lattice therapy.
* Patients with hematologic malignancies including lymphoma and leukemia as well as primary or metastatic central nervous system (CNS) malignancies.
* Patients with a history of conditions which predispose them to increased radiation toxicity
* Patients with known contraindications to radiation therapy
* Patients with uncontrolled intercurrent illness
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 60 days post treatment
  To evaluate the efficacy of lattice therapy in patients with bulky tumors, as measured by objective response rate (ORR) at 60 days post-treatment.
Adverse Events | Up to 60 days post-treatment
  To characterize the safety profile and adverse events (AEs) of lattice therapy.

SECONDARY OUTCOMES:
Overall Survival | 12 months post treatment
  To assess overall survival (OS) following lattice therapy. Overall survival will be assessed via review of medical and vital records.
Patient-reported Quality of Life | 60 days post treatment
  To determine patient-reported quality of life outcomes after lattice therapy via the Functional Assessment of Cancer Therapy - General - 7 Item Version (FACT-G7) tool as a measure of global quality of life. This is measured on 5 point Likert-type scale ranging from 0-4. Higher scores reflect better QOL.

OTHER OUTCOMES:
Impact of Lattice Therapy on Systemic Immune Anti-tumor Responses via analysis of peripheral blood samples. | Up to 5 days post-treatment
  Blood will be collected pre-treatment, after the last lattice fraction, and at 5 days post-lattice therapy for analysis via flow cytometry. Differences in immune anti-tumor responses be assessed between timepoints/tumor types. Increased immune anti-tumor responses after therapy compared to baseline are anticipated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No